CLINICAL TRIAL: NCT02750696
Title: Comparison of Two Combinations of Opioid and Non-opioid Analgesics for Acute Periradicular Abscess: A Randomized Clinical Trial
Brief Title: Comparison of Two Combinations of Opioid and Non-opioid Analgesics for Acute Periradicular Abscess
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Manuela Favarin Santin, PhD, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12671913.1.0000.5347
Record Dates: First submitted 2016-04-15; First posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Periapical Abscess
Keywords: Acetaminophen; Analgesia; Codeine; Drug Combinations; Endodontics; Periapical abscess; Randomized Controlled Trial; Tramadol; Visual analog scale
MeSH Terms: conditions — Periapical Abscess; Agnosia | interventions — acetaminophen, codeine drug combination; Ultracet

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Co/ Ac (Active Comparator): Codeine/acetaminophen (30 mg/500 mg) analgesic association tablets. Patients in this group received one fixed-dose oral tablet of codeine/acetaminophen (30 mg/500 mg) every 4 hours for 3 days.
  Interventions: Drug: Fixed-dose oral tablet of codeine/ acetaminophen every 4 hours for 3 days
- Tr/ Ac (Experimental): Tramadol/acetaminophen (37.5 mg/325 mg) analgesic association tablets. Patients in this group received one fixed-dose oral tablet of tramadol/acetaminophen (37.5 mg/325 mg) every 4 hours for 3 days.
  Interventions: Drug: Fixed-dose oral tablet of tramadol/ acetaminophen every 4 hours for 3 days

INTERVENTIONS:
Drug: Fixed-dose oral tablet of codeine/ acetaminophen every 4 hours for 3 days — Patients in this group received opioid/ non-opioid analgesic combination.
  Other Names: Codeine/ Acetaminophen (Co/Ac)
  Arms: Co/ Ac
Drug: Fixed-dose oral tablet of tramadol/ acetaminophen every 4 hours for 3 days — Patients in this group received opioid/ non-opioid analgesic combination.
  Other Names: Tramadol/ Acetaminophen (Tr/Ac)
  Arms: Tr/ Ac

SUMMARY:
Aim: The aim of this study was to compare the analgesic efficacy of two combinations of opioid and non-opioid analgesics for acute periradicular abscesses.

Methodology: This study included 24 patients who sought emergency care in a Brazilian dental school. The patients were randomly divided into two groups: Codeine/Acetaminophen - oral prescription of codeine (30 mg) plus acetaminophen (500 mg), every 4 h, for 3 days or Tramadol/Acetaminophen - oral prescription of tramadol hydrochloride (37.5 mg) plus acetaminophen (500 mg) on the same schedule. Patients recorded pain scores in a pain diary 6, 12, 24, 48, and 72 h after treatment, using the Visual Analogue Scale.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Acute Periradicular Abscess
* Age greater than 18 years
* Spontaneous pain greater than 40 mm measured in Visual Analogue Scale (moderate to severe pain).

Exclusion Criteria:

* Intake of analgesics or antibiotics within 4 hours prior to emergency surgery
* Allergy to the drugs used in this study
* Gastric ulcer, liver or kidney disease
* Uncontrolled diabetes mellitus or epilepsy
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Reduction of pain scores over time. | 0, 6, 12, 24, 48 and 72 h after first dose administration
  Pain scores were obtained using VAS before and after the first appointment.

SECONDARY OUTCOMES:
Frequency of additional medication | Up to 72 hours
  Registered in the pain diary by the patient.
Adverse reactions reported by patients | Up to 72 hours
  Registered in the pain diary by the patient.